CLINICAL TRIAL: NCT05884775
Title: iMatter2: An Artificial Intelligence (AI)-Driven Approach to Supercharge a Novel Digital Patient-reported Outcomes Tool for Diabetes Management
Brief Title: Novel Digital Patient-Reported Outcomes Tool for Diabetes Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-00608
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Telemedicine; Patient Reported Outcome Measures; prolyl-proline; Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iMatter2 (Experimental): All the patients within a primary care provider (PCP) randomized to the intervention will receive iMatter2.
  Interventions: Other: Mobile Health (mHealth) Patient-Reported Outcome (PRO) tool
- Usual Care (UC) (No Intervention): All patients within PCPs randomized to UC will receive standard Type 2 diabetes (T2D) care by their PCP.

INTERVENTIONS:
Other: Mobile Health (mHealth) Patient-Reported Outcome (PRO) tool — Once the program begins, the AI chatbot sends daily text messages that include the PRO questions; a link to a library of educational resources tailored to their responses and personalized motivational messages with support. Participants will also be sent links to the interactive web-based dashboard that visualizes their daily PRO and HbA1c data. PCPs will be able to view reports of patients' PRO and home A1c data through the EHR interface, which can be reviewed during visits with the patient or asynchronously to track patient PROs between visits.
  Other Names: iMatter2
  Arms: iMatter2

SUMMARY:
Investigators will conduct a hybrid type 1 effectiveness-implementation randomized controlled trial (RCT) to evaluate the effectiveness of iMatter2 versus usual care on reduction in HbA1c at 12-months (primary outcome) among patients with Type 2 diabetes (T2D).

ELIGIBILITY:
Inclusion Criteria:

PCP Group:

* Fulltime primary care provider (MD/DO, NP) practicing at the participating family health centers or faculty group practices and
* Provide care to at least five patients with a diagnosis of T2D

Patient Group:

* Have a diagnosis of T2D for ≥6 months;
* Have uncontrolled T2D defined as HbA1c >7% documented in the EHR on at least two visits in the past year;
* Fluency in English or Spanish;
* Be willing to send/receive text messages; and
* Be > 18 years of age.

Exclusion Criteria:

Patient Group:

* Refuse or are unable to provide informed consent;
* Have acute renal failure, end stage renal disease (ESRD) or evidence of dialysis, renal transplantation, or other ESRD-related services documented in the EHR;
* Have significant psychiatric comorbidity or reports of substance abuse (as documented in the EHR);
* Are pregnant or planning to become pregnant within 12 months;
* Currently participate in another T2D study; or
* Plan to discontinue care at the clinic within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C (HbA1c) | Baseline, Month 12
  HbA1c will be extracted from home A1c kits.

SECONDARY OUTCOMES:
Percentage of Patients Eligible for Participation in Trial who Enroll | Up to Month 14
Percentage of PCP Practices Eligible for Participation in Trial that Enroll | Up to Month 14
Percentage of Providers who View PRO Reports | Up to Month 14
Percentage of Patients who Respond to PRO Text Messages | Up to Month 14
Percentage of Patients who View PRO Interactive Dashboard | Up to Month 14
Mean Number of EHR Reports Viewed by Providers | Up to Month 14
Total Number of EHR Reports Viewed by Providers | Up to Month 14
Percentage of PRO Messages Responded To by Patients | Up to Month 14
Mean Number of PRO Messages Responded To by Patients | Up to Month 14
Total Number of PRO Messages Responded To by Patients | Up to Month 14
Mean Number of Reports Viewed by Patients via PRO Interactive Dashboard | Up to Month 14
Total Number of Reports Viewed by Patients via PRO Interactive Dashboard | Up to Month 14

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Schoenthaler, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD collected in this study will be available only to:
  • The research team, including the Principal Investigator, study coordinators, and personnel responsible for the support or oversight of the study